CLINICAL TRIAL: NCT01170312
Title: Arthroscopic Surgery and Platelet Rich Plasma In Rotator Cuff Tear Evaluation (A.S.P.I.R.E.): The Use of Platelet Rich Plasma Following Arthroscopic Repair of Rotator Cuff Tears, A Pilot Study
Brief Title: Arthroscopic Surgery and Platelet Rich Plasma In Rotator Cuff Tear Evaluation
Acronym: ASPIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Arthrex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRP-123
Record Dates: First submitted 2010-07-22; First posted 2010-07-27 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Rotator Cuff Tear
Keywords: Arthroscopic repair; Rotator cuff; Platelet rich plasma; Randomized; Pilot
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Autologous conditioned plasma (Active Comparator)
  Interventions: Biological: Autologous conditioned plasma (ACP)
- Normal saline (Placebo Comparator)
  Interventions: Other: Normal saline

INTERVENTIONS:
Biological: Autologous conditioned plasma (ACP) — ACP is not a drug as the patient's own blood plasma is re-injected into the surgical site.
  Other Names: Platelet rich plasma
  Arms: Autologous conditioned plasma
Other: Normal saline — Normal saline injection
  Arms: Normal saline

SUMMARY:
Rotator cuff tears are a common injury that lead to pain and loss of function for those who suffer from it. Treatment includes the use of arthroscopic surgery to return function to the patient and reduce their pain. This study is interested in a technique that has the potential to improve patient outcomes in terms of less pain and better function after their surgery. Autologous Conditioned Plasma (ACP) or Platelet Rich Plasma (PRP) is the intervention of interest, which is simply the patient's own blood that is withdrawn and spun down to obtain a high concentration of cells called platelets. Platelets release growth factors important for healing, as well as fibrin, which acts like a biological glue. The PRP is then re-injected into the shoulder at the time of surgery and again at 4 weeks. It has been shown to accelerate healing in other studies for injuries such as chronic elbow tendinopathy, but there is no randomized controlled trial that evaluates the effect of PRP in rotator cuff tears. It is on this basis that the study is being performed. Participating patients will receive either a PRP injection or a placebo (normal saline) and the effects will be compared at 2 weeks, 4 weeks, and 6 weeks based on a pain score and return to function questionnaires. The primary hypothesis for this study is that ACP compared with placebo is effective in reducing pain at the site of a rotator cuff injury that has undergone arthroscopic repair. It is expected that ACP administered during surgery and 4 weeks post-surgery will reduce 6-week pain scores compared to the placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Men or women who are between 18 and 70 years of age.
* Primary, traumatic or degenerative rotator cuff tears measuring 3 cm or less.
* Rotator cuff tears requiring arthroscopic repair within 18 months of initial diagnosis.
* Provision of informed consent.

Exclusion Criteria:

* Rotator cuff tears secondary to a fracture.
* Patients with an associated dislocation at the time of randomization.
* Rotator cuff tears that underwent prior surgical repair or revision arthroscopy.
* Non-surgical rotator cuff associated treatment in the 1 month prior to randomization including corticosteroid injection and anti-inflammatory treatment.
* Prior platelet rich plasma injection.
* Pre-existing conditions associated with upper extremity pain, including arthritis, ongoing infection, carpal tunnel syndrome, cervical neuropathy or other nerve pathology, local malignancy, and systemic disorders (e.g., uncontrolled diabetes, hypothyroidism).
* Patients with gross shoulder instability.
* Patients with an active infection.
* Patients who are pregnant or plan to become pregnant in the next 12 months.
* Patients with a pre-operative platelet count less than 125,000 and a pre-operative hemoglobin of 7.5g/dl or less.
* Likely problems with follow-up (i.e. patients with no fixed address, report a plan to move out of town, or intellectually challenged patients without adequate family support).
* Patients who do not read and speak English.
* Patients participating in another ongoing trial that would interfere with the assessment of the primary or secondary outcomes.
* Any other reason (in the judgment of the surgeon).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Pain score | 6 weeks
  To investigate the effect of ACP compared to placebo on pain scores in rotator cuff tears undergoing arthroscopic repair at 6 weeks.
  Pain severity will be measured using a Visual Analog Scale (VAS). Subjects will be asked to rate their worst pain in their shoulder for the previous 24 hours on a 100 mm vertical scale with "0" indicating no pain at all and "100" indicating the worst pain the subject can imagine.

SECONDARY OUTCOMES:
Physical function | Up to and including 6 weeks
  As measured by the Western Ontario Rotator Cuff Index (WORC), the Disabilities of the Arm, Shoulder and Hand Score (DASH), and the Constant Score, administered prior to the surgical intervention, and at 2 weeks, 4 weeks and 6 weeks post-surgery.
Revision surgery | Up to and including 6 weeks
Health utility | Up to and including 6 weeks
  As measured by the EuroQol-5 Dimensions (EQ-5D) administered prior to the surgical intervention, and at 2 weeks, 4 weeks and 6 weeks post-surgery.
Adverse events | Up to and including 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mohit Bhandari, MD, MSc, PhD, FRCSC, Principal Investigator — McMaster University
Locations (3):
- Canada (3):
  - McMaster University, Hamilton, Ontario
  - Hamilton General Hospital, Hamilton, Ontario
  - McMaster Hospital, Hamilton, Ontario

REFERENCES:
- [Background] Lopez-Vidriero E, Goulding KA, Simon DA, Sanchez M, Johnson DH. The use of platelet-rich plasma in arthroscopy and sports medicine: optimizing the healing environment. Arthroscopy. 2010 Feb;26(2):269-78. doi: 10.1016/j.arthro.2009.11.015. PMID 20141991
- [Background] Randelli PS, Arrigoni P, Cabitza P, Volpi P, Maffulli N. Autologous platelet rich plasma for arthroscopic rotator cuff repair. A pilot study. Disabil Rehabil. 2008;30(20-22):1584-9. doi: 10.1080/09638280801906081. PMID 18608363
- [Background] de Vos RJ, Weir A, van Schie HT, Bierma-Zeinstra SM, Verhaar JA, Weinans H, Tol JL. Platelet-rich plasma injection for chronic Achilles tendinopathy: a randomized controlled trial. JAMA. 2010 Jan 13;303(2):144-9. doi: 10.1001/jama.2009.1986. PMID 20068208